CLINICAL TRIAL: NCT06749899
Title: QL1706 (Iparomlimab and Tuvonralimab Injection,PD-1/ CTLA-4 Bi-specific Antibody) Combined With Chemoradiotherapy Versus Chemoradiotherapy Alone in High-Risk Locoregionally Advanced Nasopharyngeal Carcinoma：A Randomized, Controlled, Multicenter Phase III Clinical Study.
Brief Title: QL1706 (PD-1/CTLA-4 Bi-specific Antibody) and Chemoradiotherapy in Locoregionally-advanced Nasopharyngeal Carcinoma.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-409-FLK
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-12

CONDITIONS: Nasopharyngeal Cancinoma (NPC); Nasopharyngeal Cancer
Keywords: Immunotherapy; PD-1/CTLA-4 Bi-specific Antibody; Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL1706 Arm (Experimental): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. QL1706 5mg/kg will be given every 3 weeks for 3 cycles in induction chemotherapy and for 9 cycles in adjuvant chemotherapy, started on day 1 of induction chemotherapy and adjuvant chemotherapy, respectively.
  Interventions: Drug: QL1706; Drug: Gemcitabine; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy
- Chemoradiation Arm (Active Comparator): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: QL1706 — QL1706 5mg/kg will be given every 3 weeks for 3 cycles in induction chemotherapy and for 9 cycles in adjuvant chemotherapy, started on day 1 of induction chemotherapy and adjuvant chemotherapy, respectively.
  Arms: QL1706 Arm
Drug: Gemcitabine — Gemcitabine 1g/m2, d1 & 8 of every cycle, every 3 weeks for 3 cycles before radiation.
Drug: Cisplatin — Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation; Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
Radiation: Intensity-modulated radiotherapy — Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy will be given in 33 fractions.

SUMMARY:
The trial aimed to compare QL1706 combined with induction chemotherapy plus concurrent chemoradiotherapy (IC+CCRT) versus IC+CCRT alone in High-risk Locoregionally-Advanced Nasopharyngeal Carcinoma (LANPC).

DETAILED DESCRIPTION:
The trial plans to enroll patients with stage T4N1and T1-4N2-3 (AJCC 9th) locoregionally-advanced nasopharyngeal carcinoma (LANPC). Patients will be randomized in a 1:1 ratio to receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin and concurrent cisplatin-radiation or the same regimen plus QL1706 in induction chemotherapy and adjuvant chemotherapy. All patients will receive intensity-modulated radiotherapy (IMRT). QL1706 will begin on day 1 of induction chemotherapy and continue every 3 weeks for 3 cycles in induction therapy and for 9 cycles in adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 and ≤65 years
2. Patients with histologically confirmed non-keratinizing nasopharyngeal carcinoma according to WHO criteria.
3. Tumor staged as T4N1 and T1-4N2-3 (AJCC 9th)

   * Stage II: T1-3N2
   * Stage III: T1-4N3, T4N1-2
4. Eastern Cooperative Oncology Group performance score of 0-11.
5. Adequate marrow function: white blood cell count > 4 × 10⁹/Lhemoglobin >90g/L and platelet count >100×10⁹/L
6. Adequate hepatic and renal function：

   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×ULN
   * Alkaline phosphatase ≤ 2.5 × ULN
   * clearance rate ≥ 60 ml/min
7. Other laboratory and clinical criteria

   * Normal thyroid function, serum amylase and lipase, pituitary hormone levels, inflammatory markers, cardiac enzyme tests and electrocardiogram (ECG)
   * For patients aged >50 years with a history of smoking, normal pulmonary function test (PFT) results are required
   * For patients with abnormal ECG findings or a prior history of cardiovascular disease (not meeting any exclusion criteria listed in Item 8), additional assessments including myocardial function evaluation and cardiac ultrasound (echocardiography) must be performed, with results within normal limits
8. Patients must be informed of the investigational nature of this study and give written informed consent, and be willing and able to comply with the study schedule, including follow-up visits, treatment procedures, laboratory testing, and other protocol-related requirements.
9. Women of childbearing potential (WOCBP) must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug (e.g., condoms, physician-guided regular use of oral contraceptives).

Exclusion Criteria

1. Positive for hepatitis B surface antigen (HBsAg) with hepatitis B virus DNA >1×103 copies/mL, positive for anti-hepatitis C virus (HCV) antibody , positive for anti-hepatitis C virus (HCV) antibody
2. Positive for anti-HIV antibody or diagnosed with acquired immunodeficiency syndrome (AIDS).
3. Active pulmonary tuberculosis: Patients with a history of active tuberculosis within the past year should be excluded regardless of treatment status. Patients with a history of active pulmonary tuberculosis more than one year prior should also be excluded, unless they received confirmed and regular anti-tuberculosis treatment.
4. Active, known, or suspected autoimmune diseases, including but not limited to uveitis, colitis, hepatitis, hypophysitis, nephritis, vasculitis, systemic lupus erythematosus, hyperthyroidism, hypothyroidism, and asthma requiring bronchodilators. Type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) are allowed.
5. Thymic epithelial tumors (TETs), including thymoma, thymic carcinoma, and thymic neuroendocrine tumors (NETTs).
6. History of interstitial lung disease or pneumonia requiring oral or intravenous corticosteroids within the past year; use of vancomycin within the past month.
7. Ongoing chronic systemic corticosteroid therapy (equivalent to or greater than prednisone >10mg per day) or any other immunosuppressive therapy. Patients received inhale or topical corticosteroid are allowed.
8. Uncontrolled cardiac conditions, such as:

   * Heart failure with New York Heart Association (NYHA) classification ≥ Class II;
   * Unstable angina;
   * History of myocardial infarction within the past year;
   * Supraventricular or ventricular arrhythmias requiring treatment or intervention
9. Pregnant or breastfeeding women (pregnancy testing should be considered for women of childbearing potential with active sexual life)
10. History or presence of other malignancies, except for adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, and papillary thyroid carcinoma.
11. Known hypersensitivity to macromolecule protein products or any component of QL1706.
12. Active infections requiring systemic treatment within 1 week prior to enrollment.
13. Administration of live vaccines within 30 days prior to the first dose of epalurilimab-tovorolimab.
14. History of organ transplantation or hematopoietic stem cell transplantation.
15. Any other condition assessed by the investigator as potentially compromising patient safety or compliance, such as severe illnesses requiring urgent treatment (including psychiatric disorders), significantly abnormal laboratory values, or other psychological, familial, or social risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2025-05-04 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) in intention-to-treat population | 3 years
  Multiple endpoint 1: calculated from randomization to the date of locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first.
Overall survival (OS) in intention-to-treat population | 5 years
  Multiple endpoint 2: calculated from randomization to the date of death from any cause.

SECONDARY OUTCOMES:
Failure-free survival (FFS) in per-protocol population | 3 years
  calculated from randomization to the date of locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first.
Overall survival (OS) in per-protocol population | 3 years
  calculated from randomization to the date of death from any cause.
Locoregional recurrence-free survival (LRRFS) | 3 years
  calculated from randomization to the date of locoregional persistence or 1st locoregional recurrence.
Distant metastasis-free survival (DMFS) | 3 years
  calculated from randomization to the date of first distant metastasis.
Adverse events (AEs) and serious adverse events (SAEs) | 3 years
  Graded according to CTCAE V5.0.
Quality of life (QoL) | week 1, 20, 40, 64
  The change of QoL from randomization to the start of radiotherapy, the end of radiotherapy, 13-16 weeks after radiotherapy, 2 years and 3 years after randomization. The EORTC QoL questionnaire-C30 (EORTC QLQ-C30）version 3.0 will be used. This questionnaire comprises 30 questions, 24 of which are aggregated into nine multi-question scales, that is, five functioning scales (e.g., physical), three symptom scales (e.g., fatigue) and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual.
Failure-free survival (FFS) within different subgroups | 3 years
  analyses for FFS will be performed within the following subgroups: Epstein-Barr virus (EBV) DNA (≤4000copies/ml vs. >4000copies/ml), different PD-L1 expression levels, age, gender, performance status, T category, N category, and stage (III vs. IVA).
Tumor response | Every 6 weeks（the time of completion of induction chemotherapy, radiotherapy, and adjuvnt immunotherapy; from the date of enrollment until the date of the last time that tumorimaging and assessment of disease has been done, assessed up to 74 weeks)
  Evaluation of tumor response as CR, PR, SD, PD, NA by clinicians

OTHER OUTCOMES:
Correlation between pre-treatment PD-L1 expression level and FFS | 3 years
  Pre-treatment PD-L1 expression level of tumor cell is evaluated centrally by means of immunohistochemical testing.
Evaluate failure-free survival in the subgroup of plasma Epstein-Barr virus DNA level | 3 years
  Subgroup analysis
Evaluate failure-free survival in the subgroup of clinical stage | 3 years
  Subgroup analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Principal Investigator — Sun Yat-sen University
Locations (19):
- China (19):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hubei Province Cancer Hosiptal, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Tongji Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The Eye and ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute ＆ Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xiamen University, Fujian, Xiamen

IPD SHARING:
Plan to Share IPD: No
Complete de-identified patient data set will be submitted onto an online platform.

REFERENCES:
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Zhao Y, Ma Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Hao Y, Chen J, Zhang G, Qu S, Li Y, Feng W, Yang M, Liu B, Ouyang W, Liang J, Yu Z, Kang X, Xue S, Yang G, Yan W, Yang Y, Liu Z, Peng Y, Fanslow B, Huang X, Zhang L, Zhao H. First-in-human phase I/Ib study of QL1706 (PSB205), a bifunctional PD1/CTLA4 dual blocker, in patients with advanced solid tumors. J Hematol Oncol. 2023 May 8;16(1):50. doi: 10.1186/s13045-023-01445-1. PMID 37158938
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573